CLINICAL TRIAL: NCT01640652
Title: A Phase I, Single Centre, Open-label Dose-escalation Study to Assess the Safety and Immunogenicity of Three Doses of 25µg or 50 µg of Meningococcal Serogroup B Outer Membrane Vesicle Vaccine MenPF-1
Brief Title: MenPF-1 - A New Vaccine Against Meningococcal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011/06
Record Dates: First submitted 2012-05-23; First posted 2012-07-16 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2018-04

CONDITIONS: Serogroup B Meningococcal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose vaccine arm (Experimental): To investigate safety, tolerability and immunogenicity of 25 µg of the serogroup B meningococcal protein vaccine MenPF-1 in healthy adults aged 18 to 50 years of age when given three doses of vaccine with 8 weeks interval.
  Interventions: Biological: MenPF-1.
- High dose vaccine arm (Experimental): To investigate safety, tolerability and immunogenicity of 50 µg of the serogroup B meningococcal protein vaccine MenPF-1 in healthy adults aged 18 to 50 years of age when given three doses of vaccine with 8 weeks interval.
  Interventions: Biological: MenPF-1.

INTERVENTIONS:
Biological: MenPF-1. — A new vaccine against meningococcal disease.

SUMMARY:
In this study the investigators are testing a new vaccine against Neisseria meningitidis, the leading infective cause of childhood death in the UK. This bug (also known as meningococcus) can infect the lining of the brain (meningitis) or the blood stream (septicaemia) and can affect all ages, but especially children, adolescents and young adults.

The bug is classified into different groups based on its outer capsule (or shell), and this study will test a new vaccine to protect against group B meningococcus (MenB) disease, which is the most common type in the UK.

Vaccines are given to prepare the immune system to fight an infection. Vaccines work by stimulating the immune system to produce specialised proteins (called antibodies) and white blood cells designed to kill the bug later in life if needed.

Vaccines against other types of meningococcus have been developed and saved many lives. However MenB is different because its outer capsule does not stimulate the immune system very effectively. There is therefore no broadly effective vaccine against MenB disease.

DETAILED DESCRIPTION:
The vaccine the investigators are testing in this study is known as MenPF-1, and uses two bacterial proteins called PorA and FetA. PorA works to move particles across the bacterial cell wall, and FetA is needed to bind to iron that the bacteria need in order to grow. These proteins are found on almost all meningococcal bugs so they are an excellent target for the immune system, and it is thought that they could be the key to developing a new vaccine against MenB disease.

MenPF-1 is a type of vaccine known as an Outer Membrane Vesicle (OMV) vaccine. This means that it has been produced from 'blebs' of the meningococcal bug's outer membrane, released by the meningococcus both during natural infection and in the laboratory. These outer membrane vesicles contain the PorA and FetA proteins, so can be used to make vaccines. The techniques used to produce the OMVs to make MenPF-1 are the same as those used in other very similar safe and effective vaccines. The MenB strain that the investigators use naturally produces PorA protein, and has been genetically modified to produce increased amounts of FetA for the OMV vaccine.

MenPF-1 contains:

* Many proteins, but especially PorA and FetA
* Aluminium, which is safe and commonly used in many vaccines to better activate the immune system
* Sugar and water for injection

It is worth noting that the vaccine product MenPF-1 is designed to work against MenB and, even if successful, would not protect against all forms of meningitis. Also, it is not a live vaccine and therefore cannot cause a meningitis infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Aged between 18 and 50 years
* In good health as determined by medical history, physical examination and clinical judgment of the investigators
* (Females) Willing to use effective contraception (such as the oral contraceptive pill, contraceptive implant or barrier methods) from one month prior and for the duration of the study
* Able to attend the scheduled visits and to comply with all study procedures, including internet access for the recording of diary cards
* Willing to allow his or her General Practitioner and/or Consultant, if appropriate, to be notified of participation in the study
* Confirmation from GP that they are aware of the inclusion and exclusion criteria and are satisfied from their knowledge of the volunteer that they are suitable to enrol

Exclusion Criteria:

* History of significant organ/system disease that could interfere with trial conduct or completion
* Have any known or suspected impairment or alteration of immune function
* Study significant abnormalities on screening investigations at the discretion of an Investigator
* Receipt of a live vaccine within 4 weeks prior to vaccination or a killed vaccine within 7 days prior to vaccination
* Plan to receive any vaccine other than the study vaccine within 4 weeks following vaccination
* Scheduled procedures requiring general anaesthesia during the study
* Participant who is terminally ill
* Receipt of immunoglobulin or any blood product transfusion within 3 months of study start
* Participation in another research study involving an investigational product in the past 12 weeks, or are planning to do so within the 20 weeks of this study
* Previously having received a meningococcal B vaccine of any kind
* Previous occurrence of disease caused by N. meningitidis
* Inability, in the opinion of the Investigator, to comply with all study requirements
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Any other significant disease or disorder which, in the opinion of the Investigator, may

  * Put the participants at risk because of participation in the study
  * Influence the result of the study
  * Impair the participant's ability to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
To investigate safety and tolerability of 25 µg or 50 µg of the serogroup B meningococcal protein vaccine MenPF-1 | 20 weeks
  This will be measured by the recording and assessment of the following local and systemic adverse events following administration of each vaccine dose:
  1. Tenderness and pain at the injection site
  2. Induration
  3. Redness
  4. Swelling
  5. Headache
  6. Malaise
  7. Myalgia
  8. Nausea and/or vomiting
  9. Fever
  10. Blood parameters
  11. Any unsolicited symptom(s) not listed above

SECONDARY OUTCOMES:
Immunogenicity | 20 weeks
  Immunological assays to study the immune responses to vaccines, including:
  1. Serum bactericidal antibody (SBA) assay.
  2. Antibody concentration against vaccine antigens.
  3. Quantification of circulating vaccine-induced B-cells.
  4. Quantification of vaccine-induced, antigen specific T-cell responses and associated cytokine production.
  5. Serum opsonophagocytic activity.
  6. Gene expression profile after immunization and DNA storage for investigation of the genetic associations with the immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, PhD, Principal Investigator — Oxford Vaccine Group
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Green CA, Sande CJ, de Lara C, Thompson AJ, Silva-Reyes L, Napolitano F, Pierantoni A, Capone S, Vitelli A, Klenerman P, Pollard AJ. Humoral and cellular immunity to RSV in infants, children and adults. Vaccine. 2018 Oct 1;36(41):6183-6190. doi: 10.1016/j.vaccine.2018.08.056. Epub 2018 Aug 31. PMID 30177258
- [Result] Marsay L, Dold C, Green CA, Rollier CS, Norheim G, Sadarangani M, Shanyinde M, Brehony C, Thompson AJ, Sanders H, Chan H, Haworth K, Derrick JP, Feavers IM, Maiden MC, Pollard AJ. A novel meningococcal outer membrane vesicle vaccine with constitutive expression of FetA: A phase I clinical trial. J Infect. 2015 Sep;71(3):326-37. doi: 10.1016/j.jinf.2015.05.006. Epub 2015 May 15. PMID 25982025
- See also: OVG website — http://www.ovg.ox.ac.uk/
- See also: MenPF-1 - A New Vaccine Against Meningococcal Disease — https://clinicaltrials.gov/study/NCT01640652?locStr=Oxford,%20UK&country=United%20Kingdom&state=England&city=Oxford&distance=50&term=nct01640652&cond=meningitis&rank=1
- See also: Humoral and cellular immunity to RSV in infants, children and adults — https://pubmed.ncbi.nlm.nih.gov/30177258/
- See also: A novel meningococcal outer membrane vesicle vaccine with constitutive expression of FetA: A phase I clinical trial — https://pubmed.ncbi.nlm.nih.gov/25982025/